CLINICAL TRIAL: NCT03490305
Title: Exploratory Laparotomy Following Penetrating Abdominal Injuries From the Battle of Mosul: a Cohort Study From a Referral Hospital in Erbil, Kurdistan Region in Iraq
Brief Title: Penetrating Abdominal Injuries From the Battle of Mosul
Acronym: Exlap
Status: Completed | Type: Observational
Sponsor: Vrinnevi Hospital (Other)
Collaborators: Emergency Hospital, Erbil, Iraq (Unknown); Karolinska Institutet (Other); Center for Disaster Medicine and Traumatology, Linköping University (Unknown)
Responsible Party: Principal Investigator, Måns Muhrbeck, MD, Vrinnevi Hospital
Other Study IDs: ExlapErbil
Record Dates: First submitted 2018-03-22; First posted 2018-04-06 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Penetrating Abdominal Trauma; War Injury
Keywords: War injury; Penetrating abdominal trauma; Exploratory laparotomy; Improvised explosive device; Mosul
MeSH Terms: interventions — Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combatants: Men 16-50 years old or combatants by own admission.
  Interventions: Procedure: Exploratory laparotomy
- Civilians: Children <16 years, all women and men ≥50 years.
  Interventions: Procedure: Exploratory laparotomy

INTERVENTIONS:
Procedure: Exploratory laparotomy — Findings and procedures done at exploratory laparotomy

SUMMARY:
The battle of Mosul was characterized by the use of improvised explosive devices, human shields and suicide bombers in an urban setting. It is unclear whether this type of warfare cause more extensive abdominal injuries to civilians than combatants. All patients admitted with penetrating abdominal injury subjected to an exploratory laparotomy at Emergency Hospital, Erbil, between October 17, 2016 and July 16, 2017 will be included. Differences in demographics, injury mechanism, time since injury, clinical status on arrival, intraoperative findings, postoperative complications and outcome will be studied.

DETAILED DESCRIPTION:
Study Rationale The battle of Mosul was characterized by the use of improvised explosive devices, human shields and suicide bombers in an urban setting. It is unclear whether this type of warfare cause more extensive abdominal injuries to civilians than combatants. Understanding of the correlation between the severity of abdominal injuries, type of warfare and population affected is of importance when planning for surgical care in a conflict setting.

Aim To assess whether civilians obtain more extensive abdominal injuries than combatants in an urban battle characterized by the use of indiscriminate weapons.

Study Design An observational retrospective cohort study with longitudinal data collection.

All patients admitted with penetrating abdominal injury subjected to an exploratory laparotomy at Emergency Hospital, Erbil, between October 17, 2016 and July 16, 2017 will be included. Differences in demographics, injury mechanism, time since injury, clinical status on arrival, intraoperative findings, postoperative complications and outcome will be analysed.

Primary Objective Differences in injury mechanism, organs injured, surgical treatment given, postoperative complications and outcome between civilians and combatants.

Secondary Objectives Differences in surgical treatment given, postoperative complications and outcome between patients with prior surgical treatment of their injury and patients without prior surgical treatment.

Differences in surgical treatment given, postoperative complications and outcome between patients who receive surgical treatment less than 24 hours from injury and patients who receive surgical treatment more than 24 hours from injury will be analysed.

Statistical methods Differences between groups will be analysed using t-test and regression models.

ELIGIBILITY:
Inclusion Criteria (all must be fulfilled):

* Penetrating abdominal injury
* Subjected to an exploratory laparotomy at Emergency Hospital, Erbil, Iraq
* Between October 17, 2016 and July 16, 2017

Exclusion Criteria (all must be fulfilled):

* Patients who received treatment several times will only be counted as one patient
* Between October 17, 2016 and July 16, 2017

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted with penetrating abdominal injury subjected to an exploratory laparotomy at Emergency Hospital, Erbil, between October 17, 2016 and July 16, 2017 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Differences in injury mechanism, organs injured, surgical treatment given, postoperative complications and outcome between civilians and combatants. | an average of 3 weeks

SECONDARY OUTCOMES:
Differences in surgical treatment given, postoperative complications and outcome between patients with prior surgical treatment of their injury and patients without prior surgical treatment. | an average of 3 weeks
Differences in surgical treatment given, postoperative complications and outcome between patients who receive surgical treatment less than 24 hours from injury and patients who receive surgical treatment more than 24 hours from injury will be analysed. | an average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johan von Schreeb, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Emergency Hospital, Erbil, Kurdistan, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nassoura Z, Hajj H, Dajani O, Jabbour N, Ismail M, Tarazi T, Khoury G, Najjar F. Trauma management in a war zone: the Lebanese war experience. J Trauma. 1991 Dec;31(12):1596-9. doi: 10.1097/00005373-199112000-00005. PMID 1749028
- [Background] Coupland RM, Samnegaard HO. Effect of type and transfer of conventional weapons on civilian injuries: retrospective analysis of prospective data from Red Cross hospitals. BMJ. 1999 Aug 14;319(7207):410-2. doi: 10.1136/bmj.319.7207.410. PMID 10445921
- [Background] Sikic N, Korac Z, Krajacic I, Zunic J. War abdominal trauma: usefulness of Penetrating Abdominal Trauma Index, Injury Severity Score, and number of injured abdominal organs as predictive factors. Mil Med. 2001 Mar;166(3):226-30. PMID 11263024
- [Background] Cairns BA, Oller DW, Meyer AA, Napolitano LM, Rutledge R, Baker CC. Management and outcome of abdominal shotgun wounds. Trauma score and the role of exploratory laparotomy. Ann Surg. 1995 Mar;221(3):272-7. doi: 10.1097/00000658-199503000-00009. PMID 7717780
- [Derived] Muhrbeck M, Egelko A, Haweizy RM, von Schreeb J, Alga A. Exploratory laparotomy during the battle of Mosul, 2016-2017: results from a tertiary civilian hospital in Erbil, Iraqi Kurdistan. BMC Emerg Med. 2023 Sep 23;23(1):113. doi: 10.1186/s12873-023-00882-y. PMID 37741988

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03490305/Prot_SAP_000.pdf